CLINICAL TRIAL: NCT01432561
Title: Food-Effect on Bioavailability of Cystagon™ in Normal, Healthy Adults
Brief Title: Study in Healthy Adults to Determine the Effect That Food Has on the Absorption and Delivery of the Drug Cystagon™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Raptor Pharmaceuticals Corp. (Industry)
Responsible Party: Principal Investigator, Ranjan Dohil, Principal Investigator, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 111011
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-09

CONDITIONS: Cystinosis; Nephropathic Cystinosis
Keywords: Lysosomal Storage Diseases; Metabolic Diseases; Metabolism, Inborn Errors
MeSH Terms: conditions — Cystinosis; Lysosomal Storage Diseases; Metabolic Diseases; Metabolism, Inborn Errors | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cysteamine bitartrate (Experimental): Cysteamine bitartrate, 500mg once a day, three days.
  Interventions: Drug: Cysteamine bitartrate

INTERVENTIONS:
Drug: Cysteamine bitartrate — 500 mg total, single dose taken orally on visits 2, 3 & 4 which must occur within a 14 day period.
  Other Names: Cystagon; Cysteamine

SUMMARY:
In order to meet FDA standards of safety and efficacy reporting for most new drugs, food-effect bioavailability (the impact that the presence of food in the digestive tract has on the rate and extent at which a drug is absorbed into the bloodstream and delivered to the site of action) must be collected. Cystagon™ is an FDA approved drug for the treatment of the rare disease cystinosis that became available in 1994, but there is inadequate knowledge of the food-effect on this drug's bioavailability. This study aims to investigate how food affects the absorption of Cystagon™ into the bloodstream of normal healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, smoker (no more than 25 cigarettes daily) or non-smoker, 18 years of age and older, with BMI > 18 and < 30.0.
2. Females of childbearing potential who are sexually active must be willing to use two forms of contraceptive methods throughout the study and for 14days after the last study drug administration.
3. Minimum weight of 50 kg.
4. Good health, defined as not having history of any chronic illness and not requiring any regular medication/therapy.
5. Must swallow tablets on a regular basis.

Exclusion Criteria:

1. Evidence of Helicobacter pylori infection, presently, or within the last year.
2. Subjects with known hypersensitivity to cysteamine.
3. History, currently or within the past 3 months, of the following conditions:

   * Pancreatitis
   * Inflammatory bowel disease
   * Malabsorption
   * Severe liver disease
   * Unstable heart disease, e.g., myocardial infarction, heart failure, arrhythmias.
   * Unstable diabetes mellitus
   * Any bleeding disorder.
   * Zollinger-Ellison syndrome
   * Malignant disease
4. Subjects whom may be pregnant or have health issues that make it unsafe for them participate, or whose concomitant medical problems preclude them from committing to the study schedule.
5. Use of an investigational drug within 30 days (or 90 days for biologics) prior to dosing.
6. Use of prescription medication within 14 days prior to the first dosing;
7. Use over-the-counter products including natural health products (e.g. food supplements and herbal supplements) within 7 days prior to the first dosing.
8. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to dosing.
9. Hemoglobin <13.5 g/dL (males) and <12.0 g/dL (females) and hematocrit <41.0% (males) and <36.0% (females) at screening.
10. Breast-feeding subject.
11. Immunization with a live attenuated vaccine 1 month prior to dosing or planned vaccination during the course of the study.
12. Presence of fever (body temperature >37.6°C) (e.g. a fever associated with a symptomatic viral or bacterial infection) within 2 weeks prior to dosing.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjan Dohil, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego Center for Clinical Research Services (CCR), La Jolla, California, United States

REFERENCES:
- [Background] Gahl WA, Thoene JG, Schneider JA. Cystinosis. N Engl J Med. 2002 Jul 11;347(2):111-21. doi: 10.1056/NEJMra020552. No abstract available. PMID 12110740
- [Background] Gahl WA, Reed GF, Thoene JG, Schulman JD, Rizzo WB, Jonas AJ, Denman DW, Schlesselman JJ, Corden BJ, Schneider JA. Cysteamine therapy for children with nephropathic cystinosis. N Engl J Med. 1987 Apr 16;316(16):971-7. doi: 10.1056/NEJM198704163161602. PMID 3550461
- [Background] Markello TC, Bernardini IM, Gahl WA. Improved renal function in children with cystinosis treated with cysteamine. N Engl J Med. 1993 Apr 22;328(16):1157-62. doi: 10.1056/NEJM199304223281604. PMID 8455682
- [Background] Smolin LA, Clark KF, Thoene JG, Gahl WA, Schneider JA. A comparison of the effectiveness of cysteamine and phosphocysteamine in elevating plasma cysteamine concentration and decreasing leukocyte free cystine in nephropathic cystinosis. Pediatr Res. 1988 Jun;23(6):616-20. doi: 10.1203/00006450-198806000-00018. PMID 3393396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 09/19/2011 - 11/21/2012 Recruitment Locations: medical centers
Pre-assignment Details: Screening for liver function and H pylori infection and brief medical history in order to determine if all inclusion and exclusion criteria were met. One enrollee met all inclusion criteria but clinical lab test revealed presence of H Pylori, an exclusion factor. Two enrollees withdrew from the trial prior to assignment due to scheduling conflicts.
Groups:
- Cysteamine Bitartrate: Cysteamine bitartrate, 500mg once a day, three days.
  Cysteamine bitartrate : 500 mg total, single dose taken orally on visits 2, 3 & 4 which must occur within a 14 day period.
Period: Overall Study
Arm/Group | Cysteamine Bitartrate
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Cysteamine Absorption: Area Under the Plasma Concentration Curve (AUC)
Description: Subjects were randomized to one of two possible treatment sequences using block randomization: Sequence 1 - fasted, high-fat, high-protein or Sequence 2 - high-protein, high-fat, fasted. Sequence assignment determined the treatment condition corresponding to Period I, II & III visits.
Time Frame: 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180 minutes, and 3.5, 4, 4.5, 5, 6 hours post-dose
Measure: Mean (Standard Deviation); unit: min*uM
Groups:
- Cysteamine Bitartrate: Cysteamine bitartrate : 500 mg total, single dose taken orally on visits 2, 3 & 4
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 8
min*uM
  Fasted | 3618 (372)
  Fed High-Fat/Calorie | 2799 (405)
  Fed High-Protein | 2457 (353)
Statistical Analysis 1: Comparison: Cysteamine Bitartrate; High-fat/calorie compared to fasted condition; Test type: Superiority or Other; p = .04, ANOVA
Statistical Analysis 2: Comparison: Cysteamine Bitartrate; High-protein compared to fasted condition; Test type: Superiority or Other; p = .005, ANOVA

2. Primary Outcome: Peak Plasma Cysteamine Concentration (Cmax)
Description: as for outcome 1
Time Frame: 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180 minutes, and 3.5, 4, 4.5, 5, 6 hours post-dose
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 8
uM
  Fasted | 26.3 (3.5)
  Fed High-Fat/Calorie | 22.4 (5.6)
  Fed High-Protein | 17.2 (2.6)
Statistical Analysis 1: Comparison: Cysteamine Bitartrate; High-fat/calorie compared to fasted condition; Test type: Superiority or Other; p = .16, ANOVA
Statistical Analysis 2: Comparison: Cysteamine Bitartrate; High-protein compared to fasted condition; Test type: Superiority or Other; p = .036, ANOVA

3. Primary Outcome: Time to Peak Plasma Cysteamine Concentration (Tmax)
Description: as for outcome 1
Time Frame: 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180 minutes, and 3.5, 4, 4.5, 5, 6 hours post-dose
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cysteamine Bitartrate
Number analyzed (Participants) | 8
minutes
  Fasted | 71.2 (12.9)
  Fed High-Fat/Calorie | 106.9 (28.8)
  Fed High-Protein | 120 (23.4)
Statistical Analysis 1: Comparison: Cysteamine Bitartrate; Fed high-fat/calorie compared to fasted condition; Test type: Superiority or Other; p = .30, Non-parametric Hodges-Lehmann method
Statistical Analysis 2: Comparison: Cysteamine Bitartrate; High-protein compared to fasted condition; Test type: Superiority or Other; p = .05, Non-parametric Hodges-Lehmann method

ADVERSE EVENTS:
Time Frame: Adverse event data collected beginning date of enrollment and continuing to study withdrawal/termination or up to 7 days after last study visit, as applicable. Total duration of data collection varied among the subjects based on clinic scheduling.
Description: At study visits, subjects queried at specified intervals before and after drug administration (t=0, 30, 60, 90, 120 and 180 minutes) via a brief survey. Spontaneous A.E. observed and noted also.
  Between study visits, A.E.'s as reported by participants at the beginning of each study visit and 7 days after the final study visit were noted .
Arm/Group | Cysteamine Bitartrate
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cysteamine Bitartrate (N=8)
Nausea (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No